CLINICAL TRIAL: NCT00966485
Title: Dose-related Effect of Aspirin on Laboratory-defined Acetylsalicylic Acid Resistance and Clinical Outcome After Coronary Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Kojuri J, shiraz University of medical sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 84-2230
Record Dates: First submitted 2009-08-24; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Stenting
Keywords: ASA resistance; coronary stenting; platelet function; laboratory ASA resistance; MACE; Positive SPECT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 80 mg ASA dose (Active Comparator): 6 months post stent on 80 mg ASA
  Interventions: Drug: 80 mg ASA dosing
- 500 mg ASA dose (Active Comparator): 6 months posr stent on ASA alone
  Interventions: Drug: 500 mg ASA dosing

INTERVENTIONS:
Drug: 80 mg ASA dosing
  Arms: 80 mg ASA dose
Drug: 500 mg ASA dosing
  Arms: 500 mg ASA dose

SUMMARY:
The investigators prospectively studied the effect of aspirin on platelet function in 106 stable outpatients 6 months after successful percutaneous coronary angioplasty. Participants were randomized in a double-blind, double-crossover study (80 or 500 mg per day for 6 months).T

DETAILED DESCRIPTION:
Background:

Acetylsalicylic acid (aspirin) is widely used in the secondary prevention of coronary artery disease. There is controversy regarding the prevalence of aspirin resistance in patients with coronary artery disease and the effect of dose on resistance. Our primary aims were to determine the degree of platelet responsiveness to aspirin, and to study the influence of dose on platelet inhibition and clinical outcomes after coronary stenting.

ELIGIBILITY:
Inclusion Criteria:

* 6 months post stent without complication

Exclusion Criteria:

* subacute stent thrombosis
* unable to discontinue plavix
* dont accept to participate
* contraindication for ASA use

Ages: 40 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
laboratory ASA resistance | 6 months

SECONDARY OUTCOMES:
major adverse cardiac events and positive cardiac scan for ischemia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: javad kojuri, M.D., Study Chair — Shiraz University of Medical Sciences
Locations (1):
- Namazi hospital, Shiraz, Fars, Iran